CLINICAL TRIAL: NCT00807664
Title: Clinical Assessment of Biatain Ag Dressings Compared to Biatain Dressings in the Treatment of Leg Ulcers
Brief Title: Biatain Ag vs Biatain in the Treament of Leg Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FR008WS
Record Dates: First submitted 2008-12-11; First posted 2008-12-12 (Estimated); Results first posted 2017-12-11 (Actual); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Leg Ulcers
MeSH Terms: conditions — Leg Ulcer

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Biatain Ag dressing
  Interventions: Device: Biatain Ag
- 2 (Active Comparator): Biatain dressing
  Interventions: Device: Biatain

INTERVENTIONS:
Device: Biatain Ag — Biatain Ag non adhesive ( ColoplastA/S), a polyurethane permeable backing film with an added silver complex, size 15X15. The product is CE marked
  Arms: 1
Device: Biatain — A standard polyurethane foam dressing Biatain non adhesive permeable backing film, size15X15 cm. the product is CE marked
  Arms: 2

SUMMARY:
the objective of this investigation is to demonstrate the effect of the foam dressing Biatain Ag, compared to Biatain foam dressing( a product which is similar but does not contain a silver complex, in the healing of leg ulcers that had failed to heal despite appropriate therapy

ELIGIBILITY:
Inclusion Criteria:

* • Patients over 18 who have given written informed consent

  * Patients with a venous or predominantly venous leg ulcer (ankle-brachial index > 0.8) that is between 2 cm and 13 cm in all directions
  * Patients with a moderately or severely exudating leg ulcer in the phase of debridement or formation of granulation tissue
  * Patients with a leg ulcer that is not healing properly despite suitable and well-conducted local treatment in the four weeks prior to inclusion
  * Patients with a leg ulcer that has been treated with appropriate compression in the four weeks prior to inclusion
  * Patients who are available for monitoring for at least 10 weeks

Exclusion Criteria:

* • Patients whose leg ulcers are clinically infected (including erysipelas and cellulitis of the skin around the ulcer) requiring systemic antibiotic treatment

  * Patients who have undergone surgery on the saphenous trunk within the two months prior to inclusion
  * Patients whose leg ulcer being considered for the study has been treated with local antibiotics or antiseptics incl. dressings containing antibiotics or antiseptics in the four weeks prior to inclusion
  * Patients who have been taking systemic antibiotics in the two weeks prior to inclusion
  * Patients who have been taking systemic corticoids or cytostatics within the three months prior to inclusion
  * Patients with unbalanced diabetes at the discretion of the investigator
  * Patients with a known allergy to one of the components in Biatain Argent® or Biatain
  * Patients who are already taking part in another clinical study
  * Patients who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2008-12; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients could be in-patients, out-patients attending hospital clinics specialising in phlebo-angiology, dermatology or vascular surgery, or patients being treated in a non-hospital setting
Groups:
- Biatain Ag Wound Dressing: Biatain Ag wound dressing, is a foam wound dressing including hydro-activated silver
- Biatain Wound Dressing: Biatain dressing is a foam wound dressing
Period: Overall Study
Arm/Group | Biatain Ag Wound Dressing | Biatain Wound Dressing
Started | 88 | 94
Completed | 77 | 75
Not Completed | 11 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Biatain Ag Wound Dressing | Biatain Wound Dressing | Total
Number analyzed (Participants) | 88 | 94 | 182
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 25 | 43
  >=65 years | 70 | 69 | 139
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.1 (11.8) | 72.1 (12.4) | 73.5 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 44 | 98
  Male | 34 | 50 | 84
Region of Enrollment [Count of Participants; unit: Participants]
  France | 38 | 38 | 76
  Germany | 25 | 27 | 52
  Belgium | 3 | 1 | 4
  Denmark | 19 | 24 | 43
  United Kingdom | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change of the Leg Ulcer Area Measured by Planimetry at Week 6 Compared to the Ulcer Area at Baseline
Description: The measure of the ulcer was to measure its greatest lenght and width with these two axes being at right angles. An average of three measurements was to calculated the area of the ulcer by the equation:
  Area= Lenght *Width * pi [3.142] / 4
  All planimetry records (using double-sided tracing paper) were centrally assessed and read by a blinded person not aware of which treatment that was used.
Time Frame: Day 0 to Day 42
Population: A total of 182 subjects were randomised in the study (safety analysis set), however one patient was in systemic antibiotic treatment and was erroneously enrolled, hence the ITT analysis set comprised 181 subjects.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Biatain Ag Wound Dressing | Biatain Wound Dressing
Number analyzed (Participants) | 87 | 94
Percentage change | -41.5 (38.8) | -35.0 (44.9)

2. Secondary Outcome: Percentage Change of the Leg Ulcer Area Measured by Planimetry at Week 10 Compared to the Ulcer Area at Baseline
Description: as for outcome 1
Time Frame: Day 0 to Day 70
Population: ITT (ANCOVA) - LOCF was applied for subjects not having a value at visit 3 but a value at visit 2 for the ulcer area
Measure: Mean (95% Confidence Interval); unit: Percentage change
Groups:
- Biatain Dressing: Biatain dressing is a foam wound dressing
Arm/Group | Biatain Ag Wound Dressing | Biatain Dressing
Number analyzed (Participants) | 87 | 94
Percentage change | -59.7 [-78.8 to -40.6] | -46.1 [-65.4 to -26.8]

3. Secondary Outcome: Total Number of Adverse Events
Time Frame: Day 0 to Day 70
Measure: Number; unit: Adverse Event
Arm/Group | Biatain Ag Wound Dressing | Biatain Dressing
Number analyzed (Participants) | 87 | 94
Adverse Event
  Mild, not related | 3 | 2
  mild, possibly related | 1 | 0
  Moderate, not related | 11 | 11
  moderate, possibly related | 2 | 2
  moderate, related | 1 | 0
  severe, not related | 2 | 1
  severe, possibly related | 2 | 0
  severe, related | 0 | 2
  not specified, not related | 0 | 1

ADVERSE EVENTS:
Arm/Group | Biatain Ag Wound Dressing | Biatain Wound Dressing
Serious Adverse Events (participants affected / at risk) | 5/88 | 7/94
Other Adverse Events (participants affected / at risk) | 4/88 | 2/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Biatain Ag Wound Dressing (N=88) | Biatain Wound Dressing (N=94)
Fall (Social circumstances) | 0 (0) | 1 (1) — Unlikely related to device
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Unlikely related to device
cardiac decompression (Cardiac disorders) | 0 (0) | 1 (1) — left-complete arrythmia by artrial fibrillation. Unlikely related to device
Recurrance opposite leg mlum perforans pedis infection (Infections and infestations) | 1 (1) | 0 (0) — Unlikely related to device
pneumoccal pneumonia hypoxemiante (Infections and infestations) | 1 (1) | 0 (0) — Unlikely related to device
Arteriopathie left lower limb (Vascular disorders) | 1 (1) | 0 (0) — Unlikely related to device
acute pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Unlikely related to device
important pain on right leg (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Unlikely related to device
Artheriography planned (Investigations) | 0 (0) | 1 (1) — Unlikely related to device
Alteration of general state (Social circumstances) | 1 (1) | 0 (0) — Unlikely related to device
Attack of angina (Cardiac disorders) | 1 (1) | 0 (0) — Unlikely related to device
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) — Unlikely related to device. The patient died due to the cardiact arrest
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Biatain Ag Wound Dressing (N=88) | Biatain Wound Dressing (N=94)
Maceration - eczema - redness - pain of wound and peri-wound skin (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2) — Often AEs in form of maceration of the wound and peri-wound skin are reported together with redness, eczema and pain

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No